CLINICAL TRIAL: NCT03604406
Title: The Immunogenicity and Safety of Zostavax® and Shingrix® in Rheumatoid Arthritis Patients Using Abatacept
Acronym: BMS-188667
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kevin Winthrop (Other)
Collaborators: University of Alabama at Birmingham (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Kevin Winthrop, Associate Professor, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10433
Record Dates: First submitted 2018-07-05; First posted 2018-07-27 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Herpes Zoster; Inflammatory Disease; Rheumatoid Arthritis
Keywords: Shingles; abatacept; Varicella Zoster Vaccine
MeSH Terms: conditions — Herpes Zoster; Arthritis, Rheumatoid | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Varicella Zoster Vaccine (Zostavax) (Experimental): Live zoster vaccine injection will be administered as a single 0.65-mL dose subcutaneously in the deltoid region of the upper arm at the baseline visit
  Interventions: Biological: Varicella Zoster Vaccine
- Placebo Injection (Zostavax Comparator) (Placebo Comparator): Saline injection will be administered as a single 0.65-mL dose subcutaneously in the deltoid region of the upper arm at the baseline visit
  Interventions: Other: Placebo Injection
- Varicella Zoster Vaccine (Shingrix) (Experimental): Non-live zoster vaccine injection will be administered twice, 8 weeks apart, as a single 0.65-mL dose subcutaneously in the deltoid region of the upper arm at the baseline visit
  Interventions: Biological: Varicella Zoster Vaccine
- Placebo Injection (Shingrix Comparator) (Placebo Comparator): Saline injection will be administered twice, 8 weeks apart, as a single 0.65-mL dose subcutaneously in the deltoid region of the upper arm at the baseline visit
  Interventions: Other: Placebo Injection

INTERVENTIONS:
Biological: Varicella Zoster Vaccine — live-attenuated vaccine to prevent herpes zoster
  Other Names: Zostavax
  Arms: Varicella Zoster Vaccine (Zostavax)
Other: Placebo Injection — Saline solution injection
  Arms: Placebo Injection (Shingrix Comparator); Placebo Injection (Zostavax Comparator)
Biological: Varicella Zoster Vaccine — non-live vaccine to prevent herpes zoster
  Other Names: Shingrix
  Arms: Varicella Zoster Vaccine (Shingrix)

SUMMARY:
This investigator-initiated study will serve as a sub-study for the American College of Rheumatology-sponsored VERVE protocol currently funded by the NIH. This double-blinded multicenter randomized pragmatic trial is designed to determine whether Zostavax or Shingrix are safe and effective in patients with rheumatoid arthritis (RA) currently using anti-tumor necrosis factor (TNF) therapies. Inclusion/exclusion criteria for this sub-study mirror that of the parent VERVE trial with the exception of abatacept therapy being allowed. Preliminary data from the VERVE parent protocol enrolling patients using anti-TNF therapy is encouraging in that few patients experienced adverse events (56 adverse events in 50 participants, out of 140 participants in total) and that 96.2% of these adverse events were considered either mild or moderate. Importantly, there have been no instances of vaccine dissemination or zoster events to date.

DETAILED DESCRIPTION:
Recently, a live-attenuated vaccine (Zostavax®, Merck) to prevent herpes zoster (HZ) has been developed and approved for use among individuals age 50 years or older, regardless of previous HZ or varicella history. In a pivotal study of 38,456 older adults led by Dr. Michael Oxman (a co-investigator in the parent VERVE trial and this immunogenicity pilot sub-study), the vaccine reduced the incidence of HZ and postherpetic neuralgia (PHN) by > 50%.

Guidelines from the American Council on Immunization Practices (ACIP), based largely on expert opinion (given the absence of data), recommend that patients who use methotrexate or low to moderate doses of corticosteroids (up to 20mg/day prednisone) can receive this vaccination safely. However, theoretical concerns regarding the safety of live vaccine use in patients using biologic therapies have resulted in an ACIP recommendation that the vaccine is contraindicated in patients receiving such medications. Similarly, given a lack of data, the American College of Rheumatology (ACR) endorsed this contraindication in the updated ACR 2012 recommendations for biologic and non-biologic disease modifying anti-rheumatic drug (DMARD) use in RA patients (led by members of the project team for this present application).

Currently it is unknown if RA patients using biologics can safely receive these vaccines. Despite the demonstrated efficacy and safety of the zoster vaccine observed in non-RA patients, there are no prospective data critically examining the efficacy or safety of HZ vaccination in RA patients. The zoster vaccine was not given to immunosuppressed patients in the large Shingles Prevention Study (SPS); RA patients and others receiving biologics and immunosuppressive agents including glucocorticoids and DMARDs were excluded. However, this trial did show safety of the vaccine even for very elderly individuals including those older than 70 years of age and with little evidence of remaining VZV-specific cell mediated immunity (CMI). Moreover, live varicella vaccine has been safely given to children with HIV infection. Recently, the investigators used the administrative databases of a national U.S. Healthcare organization (Aetna) to conduct an observational study to examining Zostavax use in patients with RA and other rheumatic diseases (e.g. spondyloarthropathies). Among a total of 19,326 RA patients older than age 50, only 206 (1%) received zoster vaccine, suggesting that clinicians may be uncomfortable using the vaccine in RA patients. Additionally, approximately 60 vaccinated patients were using anti-TNF therapies within one month of vaccination, and no cases of HZ were reported during this time frame. Some studies suggest an elevated risk of HZ in RA patients using anti-TNF therapies, although HZ cases reported within these cohorts of anti-TNF users do not show increased dissemination or complications, suggesting that anti-TNF therapy might not necessarily increase the likelihood of VZV dissemination in such patients. Theoretically, however, with downregulation of interferon-gamma pathways associated with TNF blockade, an increase risk of HZ might be expected in such patients. Lastly, limited head-to-head data collected to date suggests abatacept might carry less risk of HZ and other opportunistic infections than does anti-TNF therapy. Given the widespread use of anti-TNF and other biologic therapies like abatacept, many RA patients and rheumatologists are unwilling to stop biologic therapy in order to receive Zostavax. This represents a missed opportunity with regard to HZ prevention. Clearly, given the high risk of HZ in the RA population, it would be highly beneficial to prospectively evaluate the safety and efficacy of this vaccine in patients using biologic therapy.

An additional non-live vaccine, the adjuvanted recombinant glycoprotein E (gE) herpes zoster (HZ) vaccine (recombinant zoster vaccine; RZV; Shingrix®), has recently been approved for healthy immunocompetent adults >50 years old by the Advisory Committee on Immunization Practices (ACIP). In pivotal trials among healthy individuals, the vaccine was more than 90% effective in all age groups studied (>50 years) with a low incidence of serious adverse events. However, the vaccine displayed a high degree of reactogenicity with 15.6% of individuals suffering grade 3 or higher systemic reactions. While these reactions were self-limited and typically resolved within several days, patients with active immune-mediated inflammatory diseases (e.g. RA) were not included in these trials. There is concern that given the potency of the AS01B adjuvant in RZV and its subsequent reactogenicity, that vaccination with RZV could result in flares of underlying inflammatory diseases. Further, it is unclear how biologic therapy affects the immunogenicity or reactogenicity of this vaccine, and it is possible the efficacy of this vaccine will not be as high in immunosuppressed populations. Given RZV is a non-live vaccine, it theoretically has advantage over the currently used live shingles vaccine in which it is contraindicated to give to patients using biologic therapy. However, before such use is recommended, the vaccine should be evaluated in such populations.

ELIGIBILITY:
Inclusion criteria include:

* be >= 50 years of age or older (for the Zostavax® sub-study only)
* be >= 18 years of age or older (for the Shingrix® sub-study only)
* be currently treated with abatacept therapy at the time of enrollment
* Eligible women must be post-menopausal (> 1 year since last menstrual period) or have a surgical history of bilateral oophorectomy or hysterectomy (for the Zostavax® sub-study only).
* Female participants of childbearing potential may be enrolled in the study if the participant (for the Shingrix® sub-study only):
* Has practiced adequate contraception for 30 days prior to vaccination; and
* Has a negative urine pregnancy test on the day of the first vaccination; and
* Has agreed to continue adequate contraception during the primary treatment period and for 2 months after completion of the vaccination series (Week 16)
* Patients must have a history of prior chicken pox (for the Zostavax® sub-study only; for patients who do not recall prior chicken pox, a positive varicella IgG serology can be used to document prior exposure)

Exclusion criteria include:

* prior Zostavax® receipt (for the Zostavax® sub-study only; the Shingrix® sub-study will allow prior Zostavax® receipt if 6 months or greater prior to enrollment)
* active contraindications to vaccination including allergy or sensitivity to gelatin or any other vaccine component
* acute illness or infection
* HIV/AIDS
* current systemic corticosteroid use (including any oral or parenteral use in the previous 28 days) [NOTE: this exclusion applies only for the Zostavax® portion of the study]
* methotrexate use > 25 mg/week
* dose of DMARDs not stable for > 30 days
* concomitant TNF antagonist use
* receiving radiation or chemotherapy for cancer treatment
* current leukemia
* lymphoma, or other cancer affecting bone marrow or lymphatic system
* cellular immunodeficiency
* current use (within the last 30 days) of anti-viral medications against the herpesvirus family
* Received any live virus vaccine within 28 days prior to study entry (Zostavax® sub-study only)
* Administration or planned administration of any live vaccine <28 days before the first study vaccination or through 28 days after the second study vaccination (Shingrix ® sub-study only)
* received any inactivated vaccine within 7 days prior to study entry (Zostavax® sub-study only)
* Received any inactivated vaccine +/- 14 days of each study injection (Shingrix ® sub-study only)
* known household contacts who may be susceptible to a live virus vaccine (e.g. pregnant women) [NOTE: this exclusion for the Zostavax® sub-study only]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2014-05-08 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in ELISPOT response from baseline to week 6, and one year post vaccination | 1) Baseline visit prior to vaccination; 2) 6 weeks post-vaccination; 3) 1 year post-vaccination
  Surrogate measures of vaccine efficacy will be performed on all patients using samples collected at baseline prior to vaccination, and subsequently at 6 weeks, and one year post vaccination. These measures will include:
  a. Frequency of VZV-specific T cells as measured by interferon-gamma ELISPOT assay.
  Changes in these outcome measures will be evaluated using geometric means and percentage increases in geometric means of (a) VZV-specific reactive lymphocytes.
Change in IgG titer from baseline to week 6, and one year post vaccination | 1) Baseline visit prior to vaccination; 2) 6 weeks post-vaccination; 3) 1 year post-vaccination
  Surrogate measures of vaccine efficacy will be performed on all patients using samples collected at baseline prior to vaccination, and subsequently at 6 weeks, and one year post vaccination. These measures will include:
  b. VZVgp-specific IgG titer as measured by ELISA
  Changes in these outcome measures will be evaluated using geometric means and percentage increases in geometric means of (b) VZV antibody titers in vaccine recipients as compared to placebo, as well as relative to baseline measures prior to vaccination.

SECONDARY OUTCOMES:
Development of Varicella Zoster Virus | Within 42 days of vaccination
  The primary adverse event of interest is development of varicella (ie zoster rash or disseminated complications of varicella) within 42 days of vaccination or any serious adverse event as defined according to standard regulatory definitions.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - St. Luke's Health System, Boise, Idaho
  - St. Paul Rheumatology, Eagan, Minnesota
  - Jayashree Sinha, MD, Clovis, New Mexico
  - Oregon Health & Science University, Portland, Oregon
  - Arthritis Associates, Hixson, Tennessee